CLINICAL TRIAL: NCT06327880
Title: A PHASE 1, RANDOMIZED, DOUBLE BLIND, SPONSOR OPEN, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF MULTIPLE ORAL DOSES OF PF-07054894 IN HEALTHY ADULT JAPANESE PARTICIPANTS
Brief Title: A Study to Learn About the Study Medicine Called PF-07054894 in People of Japanese Origin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: C4151006; 2023-509339-17-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07054894 (Experimental)
  Interventions: Drug: PF-07054894 or placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: PF-07054894 or placebo

INTERVENTIONS:
Drug: PF-07054894 or placebo — multiple oral doses of PF-07054894 for 14 days

SUMMARY:
The purpose of this clinical study is to learn about the safety and effects of the study medicine (PF-07054894) in healthy Japanese participants.

The study is seeking the following participants:

* Male or female Japanese participants aged 18 years or older. The participants should be healthy after going through some medical tests.
* Have a Body Mass Index (BMI) of 16 to 32 kilogram per meter squared; and a total body weight of more than 45 kilograms (100 pounds).
* Are willing and able to follow all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

In research, the participants in clinical studies are assigned by chance to separate groups that are given different treatments. Hence participants will be by chance assigned to receive either PF-07054894 or a harmless treatment that has no medical effect (placebo). Both these will be taken by mouth for 14 days. The total duration of the study is about 11 weeks, with a follow-up via telephone about 6 weeks after first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Japanese subjects aged 18 years or older
* Body Mass Index (BMI) of 16-32 kg/m2; and a total body weight >45 kg (100 lb)

Exclusion Criteria:

* Evidence or history of clinically significant disease or medical conditions
* Positive urine drug test or history of alcohol abuse or illicit drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE) or serious adverse events (SAE) | Screening, Baseline through study completion, an average of 11 weeks
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is defined as any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect. AEs include both SAEs and AEs.
Number of participants with clinically meaningful change from baseline in laboratory tests results | Screening, Baseline, Day 2, 7 and 14
Number of participants with clinically meaningful change from baseline in vital signs | Screening, Day 1, 2, 7, 14, and 15
  Number of participants with change from baseline in vital signs including supine blood pressure and pulse rate
Number of participants with clinically meaningful change from baseline in electrocardiogram (ECG) parameters | Screening, Day 1, 2, 7, 14 and 15
Maximal plasma concentration (Cmax) | Day 1 and 14
  The maximum observed plasma concentration (Cmax) will be observed directly from data.
Time to Maximum Plasma Concentration (Tmax) | Day 1 and 14
  Tmax will be observed directly from data
Area Under the Plasma Concentration-Time Profile From Time Zero (AUCτ) To End of Dosing Interval (AUCt) | Day 1 and 14
  AUCτ is summarized by dosing interval and day. Dosing interval is the interval τ between administration of doses of drug.
Half-life of PF-07054894 | Day 14
  terminal elimination half-life will be calculated based on the measured data

SECONDARY OUTCOMES:
Observed Accumulation Ratio (Rac) | Day 14
  Rac is calculated as, area under the curve from time zero to end of dosing interval on Day 14 (AUCtau) divided by area under the curve from time zero to end of dosing interval on Day 1 (AUCτ)
Observed Accumulation Ratio Based on Cmax (Rac,Cmax) | Day 14
  Rac Cmax is calculated as, maximum observed plasma concentration on Day 14 (Cmax) divided by maximum observed plasma concentration on Day 1 (Cmax)
Trough plasma concentrations (Ctrough) | Day 14
Apparent Volume of Distribution (Vz/F) as data permits | Day 14
  Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. VZ/F after oral dose is influenced by the fraction absorbed.
Apparent Oral Clearance (CL/F) | Day 14
  CL/F is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4151006